CLINICAL TRIAL: NCT01352754
Title: Prognosis Significance of Troponin T Elevation as Detected by Highly Sensitive Assay in Patient Undergoing Hip Fracture Surgery
Brief Title: Troponin T Elevation in Patient Undergoing Hip Fracture Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, David Rott, Consultant, Hadassah Medical Organization
Other Study IDs: 0394-HMO-CTIL
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Hip Fracture
Keywords: Hip fracture; Troponin T; myocardial infarction
MeSH Terms: conditions — Hip Fractures; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Patients undergoing hip fracture surgery are elderly and usually have co-morbidities; hence they are at risk for perioperative MI. Troponin is the gold standard for diagnosis of myocardial damage and currently the cornerstone of MI diagnosis. Perioperative troponin elevation is a poor prognosis factor. The significance of minor troponin elevation, detected by highly sensitivity troponin T assay, is unknown.

Objectives: To determine the frequency of perioperative troponin T elevation using highly sensitivity troponin T assay, and to determine the clinical significance of this elevation.

Methods: Serum Troponin T levels of patients undergoing hip fracture surgery will be tested prior to surgery 48 hrs and 72 hrs after surgery, using highly sensitivity troponin T assay.

Patients will be followed for 1 year. Primary outcomes- The number of patients with elevated troponin levels perioperatively and cardiac mortality at 3 months, 6 months and 1 year.

DETAILED DESCRIPTION:
Background and Rational

Hip fractures are an important cause of morbidity and mortality in the elderly. Surgery (i.e. total hip fracture surgery or replacement) is associated with better outcome; however these elderly patients have other comorbidities which put them at risk for non surgical perioperative complications .

Peri-operative myocardial infarction (MI) is associated with increased mortality and morbidity . Peri-operative MI currently diagnosed by presence of either symptoms or ischemic ECG changes, together with an elevated troponin level as measured by conventional assay.

The new highly sensitive troponin T (HS Tn T) assay, permitting measurement of concentrations that are lower by a factor of 10 than those measurable with conventional assays .

Research Objectives

The fundamental objective of our research is to further elucidate the magnitude and clinical relevance of minor perioperative TnT elevations.

Our specific objectives are:

A.To determine what is the frequency of HS Tn T elevation in patients undergoing hip fracture surgery.

B.To determine whether the presence of perioperative Tn T elevation using the HS assay is associated with higher mortality and morbidity.

Primary end points:

1. The number of patients with elevated HS Tn T levels postoperatively.
2. Cardiac mortality at 3 moths, 6 months and 1 year.

Secondary end points:

1. Total mortality at 3 moths, 6 months and 1 year.
2. Hospitalization for ACS and/or CHF at 3 months, 6 months and 1 year.

Methods

Patients admitted with traumatic femoral neck fracture will be recruited if surgery is planned.

Clinical evaluation for symptoms and signs of myocardial ischemia will be performed prior to surgery and 24 hrs after surgery.

Serum Tn T levels will be tested prior to surgery 48 hrs and 72 hrs after surgery, using HS Tn T assay.

ECG monitoring will be performed prior to surgery and 24 hrs after surgery. Patients will be followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years, admitted with traumatic femoral neck fracture undergoing surgery

Exclusion Criteria:

* Patients who will not undergo surgery
* Patients whom clinical singes and baseline troponin (prior to surgery) will suggest an acute myocardial infarction
* Patient younger than 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted with traumatic femoral neck fracture
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The number of patients with elevated HS Tn T levels post operatively. | One year
Cardiac mortality | one year

SECONDARY OUTCOMES:
Total mortality | One year
Any hospitlization | One year

CONTACTS AND LOCATIONS:
Overall Officials: David Rott, MD, Principal Investigator — Hadassah-Hebrew University Hospital
Locations (1):
- Hadassah hebrew university medical centers, Jerusalem, Israel